CLINICAL TRIAL: NCT04004234
Title: A Phase I/II, Open-label, Single-center Study to Evaluate the Safety and Efficacy of the Pan-immunotherapy in Subjects With Local Advanced/Metastatic Biliary Tract Cancer
Brief Title: A Phase I/II Study of the Pan-immunotherapy in Patients With Local Advanced/Metastatic BTC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-042
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Biliary Tract Cancer (BTC)
Keywords: local advanced; metastatic; anti-PD-1 antibody; Manganese; gemcitabine; cisplatin
MeSH Terms: conditions — Biliary Tract Neoplasms; Neoplasm Metastasis | interventions — manganese chloride; 130-nm albumin-bound paclitaxel; Paclitaxel; Injections; Gemcitabine; spartalizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manganese primed anti-PD-1 antibody plus nPG chemotherapy (Experimental): Subject received Manganese primed anti-PD-1 antibody, nab-paclitaxel and gemcitabine every 3 weeks until achieving a second assessable stable disease or up to a maximum of 12 cycles. Treatment continued until progressive disease, development of unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Manganese Chloride; Drug: nab-paclitaxel; Drug: Gemcitabine; Drug: anti-PD-1 antibody

INTERVENTIONS:
Drug: Manganese Chloride — Administered by inhalation at 0.2 or 0.4mg/kg/d once daily in a 3-week cycle
Drug: nab-paclitaxel — Administered intravenously, 125mg/m2/d on day1 and day8 in a 3-week cycle
  Other Names: Paclitaxel For Injection (Albumin Bound)
Drug: Gemcitabine — Administered intravenously, 1g/m2/d on day1 and day8 in a 3-week cycle
Drug: anti-PD-1 antibody — Administered intravenously, 2-4mg/kg on day 3 in a 3-week cycle
  Other Names: Anti-PD-1 monoclonal antibody; PD-1 inhibitor

SUMMARY:
Biliary tract cancer (BTC) is a rare heterogeneous collection of malignancies arising within the biliary tract, characterized by innate chemoresistance and abysmal prognosis. PD-1 blockade has been developed to a new class of cancer immunotherapy that could restore an adequate immunosurveillance against the neoplasm and enhance T-cell-mediated anticancer immune responses. Manganese has been confirmed to activate antigen-presenting cells and function as mucosal immunoadjuvants in pre-clinical studies. This open-label, phase I/II study is designed to assess the safety and efficacy of Manganese primed combined therapy of anti-PD-1 antibody and gemcitabine/cisplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old.
2. Life expectancy of at least 3 months.
3. Subjects must have Histopathological/cytological diagnosis of unresectable or recurrent /metastatic biliary tract carcinoma (intra-hepatic, extrahepatic or gall bladder).
4. Eastern Cooperative Oncology Group performance status 0-2.
5. Subjects must have at least one measurable lesion ≥ 1 cm as defined by response criteria.
6. Subjects may have received prior radiotherapy, chemotherapy, or other local ablative therapies, which completed ≥ 4 weeks prior to registration AND patient has recovered to <= grade 1 toxicity.
7. Subjects with Anti-PD-1 antibody treatment history are eligible which must be resistance.
8. Adequate organ function.
9. Participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Prior organ allograft.
4. Women who are pregnant or breastfeeding.
5. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
6. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with treatment-related adverse events (AEs) | 12 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0. AEs were considered to be treatment-related if they had started or worsened within the interval from first study drug administration until the follow-up visit.
Progression-free survival (PFS) at 6 months | 6 months
  Progression free survival (PFS) at 6 months in patients with local advanced /metastatic BTCs treated with the combined regimen. Progression will be defined clinically or on imaging as per immune related response evaluation criteria in solid tumors (RECIST V1.1) definition

SECONDARY OUTCOMES:
Disease control rate (DCR) | 12 months
  DCR is defined as the proportion of subjects who achieved a stable disease (SD), partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Object response rate (ORR) | 12 months
  ORR is defined as the proportion of subjects who achieved a partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Overall survival (OS) | 24 months
  OS time was measured from the study entry to the date of death.
Number of participants with laboratory test abnormalities | 12 months
  The laboratory tests of serum cytokines and chemokines will be performed on day 1 and 3 of each cycle, and the abnormality will be determined by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China